## The assessment of maxillary stability in Bimaxillary orthognathic patients treated by mandible-first approach versus maxilla-first approach; Randomized controlled clinical trial.

Department of Oral and Maxillofacial Surgery, Faculty of Oral & Dental Medicine, Cairo University

In partial fulfillment of the requirements for the Doctorate degree

## Submitted by:

Mohamed Hamdy Mahmoud Ismail
B.D.S 2010
M.D.S 2016
Faculty of Oral & Dental Medicine
Cairo University

16\11\2017

## Roles and responsibilities:

- 1. Ass. Prof. Dr. Niven Askar (NA)
  - Assistant Professor of Oral and Maxillofacial Surgery Cairo University
- The senior supervisor
- 2. Dr. Tarek El-Faramawi (TF)
- Lecturer Oral and Maxillofacial Surgery Cairo University
- Assistant supervisor
- 3. Dr. Mohamed Hamdy (MH)
- Assistant lecturer of Oral and Maxillofacial Surgery MSA University
- Principle Investigator

## **Consent Form**

| ation name. | |
|--------------------------------------------------------------|----|
| .ge: | |
| ddress: | |
| have approved to be enrolled in this research project and th | ne |
| esearcher has explained all the surgical procedure and its | |
| xpected outcomes and common complications that could | |
| appen and their management | |

Patient signature

Patient name:

Researcher signature